CLINICAL TRIAL: NCT02694341
Title: Bakri Ballon With or Without Abdominal Traction Stitch in Management of Uterine Bleeding in Cases of Placenta Previa
Brief Title: Bakri Balloon in Placenta Previa
Acronym: BB-ATS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants shared
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BB
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Bleeding; Placenta Previa
Keywords: Management
MeSH Terms: conditions — Hemorrhage; Placenta Previa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bakri Balloon with abdominal traction stitch (Active Comparator): bakri balloon will be inserted with abdominal traction stitch
  Interventions: Procedure: Abdominal traction stitch; Device: Bakri Balloon
- Bakri Balloon without abdominal traction stitch (Experimental): bakri balloon will be inserted with no performance of abdominal traction stitch
  Interventions: Device: Bakri Balloon

INTERVENTIONS:
Procedure: Abdominal traction stitch — Abdominal traction stitch to prevent prolapse of the Bakri balloon. A suture is tied through the uterine end shaft hole of the Bakri balloon. The other end of the suture is placed through the uterine wall. The balloon is positioned in the lower segment.The abdominal traction stitch is held by forceps and fixed, with cephalad traction applied continuously to the balloon, preventing balloon prolapse.The abdominal traction stitch is fixed by an umbilical cord clamp on the abdominal wall, preventing the suture from receding into the abdominal cavity, and, thus, maintaining the correct position of the balloon and preventing prolapse. Removal of the balloon is easy, with no resistance; the suture does not hinder balloon removal. At the time of balloon removal, the suture that was placed through the abdominal wall will traverse the intra-abdominal and intrauterine cavities, and should be kept clean.
  Arms: Bakri Balloon with abdominal traction stitch
Device: Bakri Balloon — uterine compression balloon

SUMMARY:
The Bakri intrauterine balloon can achieve haemostasis in cases of postpartum haemorrhage, including haemorrhage associated with placenta previa by compressing the lower uterine segment.

ELIGIBILITY:
Inclusion Criteria:

1. All women delivered and presented with primary atonic PPH
2. Women who accepted to participate

Exclusion Criteria:

1. Traumatic PPH as excluded by examination under anesthesia.
2. With any suspected or clinical evidence of uterine infection
3. Women diagnosed to have preeclampsia or eclampsia after delivery.
4. Women who had DM during pregnancy
5. Women with history of DVT or other thromboembolic complication
6. Women with history of rheumatic heart disease.
7. Women with coagulation defects.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percentages of failure of Bakri Balloon either rupture of balloon or slippage of balloon. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374